CLINICAL TRIAL: NCT00888680
Title: A Multinational, Multi-centre, Randomised, Double-blind, Placebo-controlled, 3-way Crossover Study in Migraine Patients, Treated With Two Doses of BGC20-1531 and Placebo
Brief Title: Double-blind, Placebo-controlled Study of BGC20-1531 in Migraine
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patients enrolled. Delay due to optimisation of drug product formulation.
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BGC20-1531-06
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Migraine
Keywords: Migraine; Headaches; Migraine headaches; Head pain
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — N-(4-(4-(5-methoxypyridin-2-yl)phenoxymethyl)-5-methylfuran-2-carbonyl)-2-methylbenzenesulfonamide; Lactose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- BGC20-1531 200 mg (Experimental)
  Interventions: Drug: BGC20-1531
- BGC20-1531 400mg (Experimental)
  Interventions: Drug: BGC20-1531
- Lactose (Placebo Comparator)
  Interventions: Drug: Lactose

INTERVENTIONS:
Drug: BGC20-1531 — BGC20-1531 administered orally
  Arms: BGC20-1531 200 mg; BGC20-1531 400mg
Drug: Lactose — Placebo administered orally
  Arms: Lactose

SUMMARY:
The study is being conducted to explore the safety and effectiveness of a new chemical entity, BGC20-1531, in subjects with a history of migraine. In this study subjects will treat a total of three migraine attacks with two different doses of BGC20-1531 and placebo, with at least one week wash out period between doses.

DETAILED DESCRIPTION:
Migraine headache is estimated to affect 10-20% of the world population and is listed by the World Health Organisation in the top 20 causes of disabling conditions, and in the top four neurological disabling conditions. The most common therapies for acute migraine are non-steroidal anti-inflammatory drugs (NSAIDs) and triptans. However, many migraine sufferers do not experience sufficient relief from these treatments or cannot tolerate their gastrointestinal, cardiovascular and other side-effects.

Prostaglandin PGE2-induced sensory nerve sensitisation, neuropeptide release and cerebral vascular dilatation is thought to underlie migraine pain, particularly via activation of the EP4 receptor subtype. BGC20-1531 is an orally available EP4 receptor antagonist which inhibits prostaglandin-induced vasodilation of cranial blood vessels via a selective blockade of EP4 receptors reducing inflammation and migraine pain. As EP4 receptors are discretely localised, the overall safety profile of EP4 receptor antagonists may be improved compared to triptans and NSAIDs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine (with or without aura) according to the criteria of the International Headache Society.
* Age at onset of migraine less than 45.0 years.
* Males and females between 18.0 and 65.0 years of age inclusive.
* Be willing and able to give written informed consent.
* For female patients, a negative pregnancy test
* Sexually active participants and their partners should be using an effective method of contraception; combined hormonal or progestogen-only methods, IUD/IUS, diaphragm/condoms with spermicide or sterilisation.
* History of 1-6 migraine attacks per month (with or without aura) in the 3 months prior to screening, with at least 48 hours freedom from headache between attacks.
* Patients receiving migraine prophylactic treatment can be enrolled, providing they are receiving only one drug for prophylaxis and the prescribed daily dose is not changed in the month prior to screening.
* Rescue medication is permitted in the study.
* Women with menstrual migraine (or who have suspected menstrual migraine or are subsequently diagnosed with menstrual migraine) may be included in the study and instructed to treat each consecutive attack with study medication (unless within the wash-out period).
* Patients who are willing and able to comply with study requirements including completion of the study diary.
* Patients who are taking prescribed medication for depression may be included providing this treatment has been stable for 3 months prior to screening and is expected to remain stable for the duration of the study.
* In the investigators opinion are suitable for inclusion in the study.

Exclusion Criteria:

* Patients with ≥15 headache days (migraine and non-migraine headaches combined) per month.
* Patients who take analgesics for any reason ≥15 days a month or triptans ≥10 days a month.
* Non-migraine headaches on more than 6 days per month.
* Patients with schizophrenia.
* Patients prescribed more than one migraine prophylaxis treatment.
* Patients receiving prophylaxis whose prescribed daily dose has changed within the month before screening.
* Patients whose prophylactic treatment is not expected to remain stable for the duration of the study.
* Patients whose prophylactic treatment has been withdrawn within the month prior to study entry.
* Patients taking ergotamine, ergotamine derivatives or ergotamine combination products.
* Any relevant abnormality on history or examination including central nervous system, psychiatric (excluding depression), respiratory, cardiovascular or metabolic dysfunction.
* Abnormal laboratory findings suggesting infectious, endocrine, malignant disease or other systemic disorder; any isolated abnormal laboratory finding considered clinically relevant by the investigator at screening.
* Subjects with clinically significant abnormalities in 12-lead electrocardiogram (ECG), blood pressure and/or pulse at screening.
* Recent or clinically significant history of drug or alcohol abuse.
* Inability to communicate well with the investigator (ie, language problem, poor mental development or impaired cerebral function).
* Participation in a clinical study of an Investigational Medicinal Product (IMP) within the 3 months up to screening.
* Patient unable to commit to participating in the clinical study for up to 8 months or patient expecting any medical interventions during that time.
* Patients taking prescribed medication for depression, whose treatment has not been stable for 3 months up to screening and is not likely to remain stable for the duration of the study.
* Female patients who are pregnant or lactating.
* Patients taking any unapproved herbal remedies for treatment of depression or migraine e.g. feverfew, St Johns Wort. (Supplementary vitamins, minerals or homeopathic remedies will be permitted provided their intake is kept constant throughout the study).
* Patients with a history of lactose intolerance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of BGC20-1531 on headache response, defined as a decrease of headache from severe or moderate to mild or none at 2 hours post-dose without the use of rescue medication. | 2 hours

SECONDARY OUTCOMES:
To evaluate the effect of BGC20-1531 on pain-freedom up to 48 hours post-dose without the use of rescue medication. | Up to 48 hours
To evaluate the effect of BGC20-1531 on headache response up to 48 hours post-dose (without the use of rescue medication). | Up to 48 hours
To evaluate the effect of BGC20-1531 on sustained headache relief and pain-freedom over a 24-hour and 48-hour period post-dose. | Up to 48 hours
To evaluate the safety of BGC20-1531. | Duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Messoud Ashina, MD, Principal Investigator — Danish Headache Center
Locations (4):
- Danish Headache Center, Glostrup Municipality, Denmark
- Norway (2):
  - Head and Neck Research Group, Oslo
  - Norwegian National Headache Centre, Trondheim
- The City of London Migraine Clinic, London, United Kingdom